CLINICAL TRIAL: NCT03410849
Title: Long-term Adverse Effects After Laparoscopic Sleeve Gastrectomy and Roux en Y Gastric Bypass (Part B)
Brief Title: Long-term Adverse Effects After Bariatric Surgery on Oesophagus Epithelium
Acronym: FUB-B
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FUB Study Oesophagus
Record Dates: First submitted 2018-01-02; First posted 2018-01-25 (Actual); Last update posted 2020-11-03 (Actual); Status verified 2020-11

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid | interventions — Gastroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric Bypass (Active Comparator): A gastroscopy will be carried out to document the presence of inflammation and metaplasia in patients after an average of 5 years after laparoscopic gastric bypass
  Interventions: Diagnostic Test: Gastroscopy
- Sleeve Gastrectomy (Active Comparator): A gastroscopy will be carried out to document the presence of inflammation and metaplasia in patients after an average of 5 years after laparoscopic sleeve gastrectomy
  Interventions: Diagnostic Test: Gastroscopy

INTERVENTIONS:
Diagnostic Test: Gastroscopy — in both arms intervention 'gastroscopy' will be carried out

SUMMARY:
The goal of this trial is to examine long-term effects of laparoscopic gastric bypass (LRYGB) and sleeve gastrectomy (LSG) on oesophageal symptoms and disease, including the presence of Barrett oesophagus ≥ 5 years post-surgery.

DETAILED DESCRIPTION:
Bariatric surgery shows impressive results in terms of weight loss and resolution of comorbidities. Still, there are questions as to the frequency of long-term adverse effects: the prevalence and causes of post-operative swallowing disorders and reflux disease are uncertain. Recently, independent study groups described a high incidence of Barrett oesophagus post LSG. Additional research is urgently needed.

The goal of this trial is to examine long-term effects of laparoscopic gastric bypass (LRYGB) and sleeve gastrectomy (LSG) on oesophageal symptoms and disease, including the presence of Barrett oesophagus ≥ 5 years post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received laparoscopic gastric bypass or laparoscopic sleeve gastrectomy ≥ 5 years ago as a primary bariatric procedure will be eligible for this study.

Exclusion Criteria:

* Patients who received laparoscopic gastric bypass or laparoscopic sleeve gastrectomy as a secondary bariatric procedure (e.g. after gastric banding),
* Patients who received a secondary bariatric operation after laparoscopic gastric bypass or laparoscopic sleeve gastrectomy( e.g. biliopancreatic diversion)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 170 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Incidence of Barrett oesophagus after bariatric surgery | 5-7 years after bariatric surgery
  incidence of Barrett oesophagus will be compared to will be compared to reference for this age

SECONDARY OUTCOMES:
Prevalence of dysphagia after bariatric surgery | 5-7 years after bariatric surgery
  Prevalence of dysphagia will be compared to will be compared to reference for this age
Prevalence of oesophageal motility disorders after bariatric surgery | 5-7 years after bariatric surgery
  Prevalence of oesophageal motility will be compared to will be compared to reference for this age

CONTACTS AND LOCATIONS:
Overall Officials: Bettina Wölnerhanssen, MD, Principal Investigator — Clinical Research St Claraspital
Locations (1):
- St Claraspital, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No